CLINICAL TRIAL: NCT07156435
Title: A Phase lb Study of Vyxeos® (Liposomal Daunorubicin and Cytarabine) in Combination With Clofarabine in Children With Relapsed/Refractory AML, ITCC-092
Brief Title: Vyxeos® With Clofarabine for Pediatric AML
Acronym: VyClo
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Princess Maxima Center for Pediatric Oncology (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITCC-092; 2020-000142-34 (EudraCT Number); 2023-508050-26 (EudraCT Number); NL72866.041.20 (Other: CCMO)
Record Dates: First submitted 2025-08-19; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Relapsed Pediatric AML; Refractory Pediatric AML
Keywords: pediatric AML; relapsed/refractory; clofarabine; liposomal daunorubicin and cytarabine
MeSH Terms: conditions — Recurrence | interventions — Liposomes; Clofarabine

STUDY DESIGN:
Intervention Model Description: Open label, non-randomized, Phase 1B dose finding study following a rolling-6 design, with a dose-escalation part followed by an expansion cohort to better characterize safety at the RP2D.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with Vyxeos®/CPX-351 in combination with clofarabine (Experimental): Treatment will consist of 2 courses. An adapted regimen is used to combine Vyxeos®/CPX-351 at a fixed dose given at day 1, 3, 5 with clofarabine at the allocated dose level given at day 2-6 in course one, and only Vyxeos®/CPX-351 in course 2.
  A maximum of 3 dose levels of clofarabine are expected to be tested in this study.
  Interventions: Drug: Vyxeos 44 MG / 100 MG Liposome Injection; Drug: Clofarabine

INTERVENTIONS:
Drug: Vyxeos 44 MG / 100 MG Liposome Injection — Vyxeos®/CPX-351 will be infused in 90 minutes on day 1, 3 and 5 only, 3 hours after the end of clofarabine (if administered on the same day).
Drug: Clofarabine — Clofarabine infusion will be given according to the assigned dose level, over 2 hours IV, daily on day 2-6 (for 5 consecutive days).

SUMMARY:
Treatment with intensive chemotherapy in AML results in approximately 70% survival in newly diagnosed patients. Prognosis at relapse is worse and is in the 30-40% range. Relapse treatment generally consists of one course of fludarabine, cytarabine and liposomal daunorubicin (FLAG-DNX), followed by a fludarabine and cytarabine course, and subsequent stem-cell transplantation. Cytarabine has been used in combination with fludarabine and cladribine, with the aim to induce synergism by increasing Ara-CTP (active cytotoxic metabolite from ara-C) accumulation, which can be seen as a surrogate marker for cytarabine induced cell-kill. Synergy with cytarabine can also be achieved with clofarabine, which is a potent inhibitor of ribonucleotide reductase, leading to a depletion of normal deoxynucleotides and subsequently to increased Ara-CTP levels. The phase IB trial ITCC020/I-BFM 2009-02 recently reported that clofarabine, replacing fludarabine in the standardly used fludarabine, cytarabine and liposomal daunorubicin (FLAG-DNX) combination regimen, showed high response rates (Overall Response Rate - ORR 68% and 80% at the recommended phase 2 dose - RP2D) in patients with refractory/relapsed AML, and was generally tolerable, with infectious complications as the main side-effect due to the immunosuppressive properties of clofarabine.

Currently DNX is unavailable, which urges the need to develop other treatment blocks. The liposomal formulation of Vyxeos®/CPX-351 may be a suitable replacement for DNX, considering the long-term side effect of cardiotoxicity due to anthracyclines which is of primary importance in younger heavily pre-treated patients. The hypothesis is that due to the liposomal formulation there is less penetrance in the cardiac muscle and hence less cardiac damage. The results in pediatric and young adult patients with relapsed/refractory AML in a COG study using Vyxeos®/CPX-351 at a RP2D of 135 U/m2 (AAML1421) showed encouraging ORR, with 70% of patients reaching CR/CRi as best response after single agent-treatment with Vyxeos®/CPX-351. Preclinical data have also demonstrated an increased Ara-CTP accumulation and cytotoxicity in cell lines, and were confirmed by tests in ex-vivo blasts from a cohort of AML patients (n=5), when cells were exposed to Vyxeos®/CPX-351 after 4 hours of incubation with fludarabine.

In this study Vyxeos®/CPX-351 was evaluated in combination with clofarabine with the aim to establish the RP2D of this combination.

ELIGIBILITY:
We will include pediatric patients ≥1 year and ≤21 years with:

* Any ≥ 2nd relapse of AML
* Refractory AML (defined as ≥ 20% blasts in the bone marrow after standard (re-) induction therapy)
* Early 1st relapse (defined as relapse within one year from initial diagnosis) of AML
* Any relapse of AML after prior allogenic HSCT
* Any relapse of AML with high risk cytogenetic characteristics (as defined in Appendix V)

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

Initial work-up:

• Complete initial work-up within 7 days prior to study entry, including bone-marrow aspiration, lumbar puncture (without intrathecal therapy)

General condition:

* Lansky play score ≥ 60 for patients <16 years of age; or Karnofsky performance status ≥ 60 for patients ≥ 16 years of age (see Appendix I for Performance scales).
* Life expectancy > 6 weeks
* The patient must have a calculated GFR ≥ 70mL/min/1.73 m2.
* Liver function: total serum bilirubin ≤ 3 mg/dl or 50 μmol/L and aspartate transaminase (AST) and alanine transaminase (ALT) ≤200 U/L
* Adequate cardiac function (defined as shortening fraction ≥28% or ejection fraction ≥50%)
* No evidence of a currently uncontrolled bacterial, viral or parasitic infection
* No evidence of a fungal infection, defined as either:

  * Pulmonary infiltrates suggestive of a fungal infection at HR-CT (within 3 weeks prior to enrollment)
  * Positive Aspergillus serum test (galactomannan), according to local laboratory practice (within 3 weeks prior to enrollment)
* No evidence of isolated extramedullary relapse, including isolated CNS-relapse
* No evidence of CNS3 or symptomatic CNS leukemia
* No Down Syndrome
* No evidence of relapsed/refractory acute promyelocytic leukemia (APL)
* No use of any anticancer therapy within 2 weeks before study entry. The patient must have recovered from all acute toxicities from any previous therapy (note: hematological toxicities do not need to be considered since the patient has overt leukemia)
* No history of prior veno-occlusive disease (VOD)
* No known hypersensitivity to cytarabine, clofarabine or liposomal daunorubicin
* No known copper metabolism deficiency, such as Wilson's disease.

Other:

* For female patients with childbearing potential, a negative test for pregnancy is to be performed before entry on study.
* Male and female patients must use a highly effective contraceptive method according to the CTFG 2014-guidelines during the study and for a minimum of 6 months after study treatment.

NL72866.041.20 / Vyxeos liposomal and Clofarabine in R/R pediatric AML - ITCC-092 Protocol version: 2.2, 08-04-2021 38 of 80

* Female patients may not breast feed during the study and for a minimum of 3 months after study treatment.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule is required; those conditions should be discussed with the patient before registration in the trial.
* Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations.

Concomitant treatments:

* Concomitant administration of any other experimental drug under investigation, or concurrent treatment with any other anti-cancer therapy other than specified in the protocol is not allowed.
* GCSF will not be used for priming and no routine GCSF support is allowed during the 1st course, except for life-threatening infections.

Additional criteria:

• At least 6 patients must be enrolled with an M3 or a WBC count >10x109/L with blasts.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-11-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose finding for combination Vyxeos® with clofarabine | 2 years
  To establish the recommended phase 2 dose of Vyxeos®/CPX-351 in combination with clofarabine in children with relapsed/refractory AML

SECONDARY OUTCOMES:
To determine the safety and tolerability of Vyxeos®/CPX-351 in combination with clofarabine by observing dose-limiting toxicities (DLTs) | 4 years
To determine the (preliminary) efficacy in terms of the hematological remission rate in these patients as determined by morphology with flow cytometric confirmation | 4 years
To describe the durability of response, including the number of patients that undergo stem- cell transplant after re-induction with this regimen | 4 years

OTHER OUTCOMES:
To describe the pharmacokinetics parameters: serum concentration of Vyxeos® components (cytarabine and daunorubicin) and metabolites | 4 years
To describe the relationship between response (ORR) and intracellular Ara-CTP accumulation | 4 years
To describe the correlation between duration of response and measurable residual disease assessed by Flow-cytometry | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: C.M. Zwaan, Prof. dr., Principal Investigator — Princess Maxima Center
Locations (13):
- St. Anna Kinderspital, Vienna, Austria
- Rigshospitalet, Copenhagen, Denmark
- Germany (5):
  - Universitätsklinikum Augsburg, Augsburg
  - Charité Berlin, Berlin
  - University Children´s Hospital III Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
- Italy (2):
  - Clinica Pediatrica Fondazione MBBM, Monza
  - Ospedale Pediatrico Bambino Gesu (OPBG), Roma
- Princess Maxima Center, Utrecht, Utrecht, Netherlands
- Spain (3):
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Vall D'Hebron, Barcelona
  - Hospital Infantil Universitario Niño Jesús, Madrid

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR